CLINICAL TRIAL: NCT00172302
Title: Can Intravenous Vitamin C Improve Skin Hyperpigmentation in Long-Term Hemodialysis Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 930105
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-05

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ascorbic Acid; Injections, Intravenous

INTERVENTIONS:
Drug: vitamin C, intravenous injection

SUMMARY:
Intravenous vitamin C may improve skin hyperpigmentation in chronic hemodialysis patients

DETAILED DESCRIPTION:
Melanogenesis is caused by enzymatic conversion of tyrosine to melanin pigments.Ascorbic acid has the ability to inhibit peroxidase and may thus inhibit melanin synthesis.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis patients

Exclusion Criteria:

* allergic to vitamin C, using steroid, etc

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-11

PRIMARY OUTCOMES:
Skin pigmentation extent

SECONDARY OUTCOMES:
blood anti-oxidant level

CONTACTS AND LOCATIONS:
Overall Officials: Kao Tze-Wah, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan